CLINICAL TRIAL: NCT03443960
Title: A Multiple-Dose, Randomized, Open-Label, Parallel Pharmacokinetic Comparison Study of TNX-102 SL (Cyclobenzaprine Hydrochloride [HCl] Sublingual Tablets) 2 x 2.8 mg Versus AMRIX® (Cyclobenzaprine HCl ER Capsules) 30 mg in Healthy Subjects Under Fasting Conditions
Brief Title: Steady-State Pharmacokinetic Comparison Study of TNX-102 SL 5.6 mg Versus AMRIX® 30 mg ER Capsules
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tonix Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TNX-CY-F106
Record Dates: First submitted 2018-02-06; First posted 2018-02-23 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — cyclobenzaprine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A (TNX-102 SL) (Experimental): 2 x TNX-102 SL (cyclobenzaprine HCl sublingual tablets) 2.8 mg once daily for 20 consecutive days
  Interventions: Drug: TNX-102 SL 5.6 mg
- Treatment B (AMRIX) (Active Comparator): 1 x AMRIX ER capsule 30 mg once daily for 20 consecutive days
  Interventions: Drug: Amrix 30 mg

INTERVENTIONS:
Drug: TNX-102 SL 5.6 mg — Subjects randomly assigned to this treatment will place 2 tablets simultaneously under the tongue until dissolved, and not to crush or chew them.
  Other Names: cyclobenzaprine HCl
  Arms: Treatment A (TNX-102 SL)
Drug: Amrix 30 mg — Subjects randomly assigned to this treatment will swallow 1 capsules with a cup of water, and not to crush or chew it.
  Other Names: cyclobenzaprine HCl
  Arms: Treatment B (AMRIX)

SUMMARY:
This will be a single center, comparative pharmacokinetic, open-label, randomized, multiple-dose, 1-period, 2-arm, parallel study of TNX-102 SL 5.6 mg (administered as 2 x 2.8 mg tablets) to AMRIX® (cyclobenzaprine hydrochloride [HCl] extended-release [ER] capsules), 30 mg.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, non-smoker, ≥18 and ≤75 years of age (Treatment A) or ≥18 and ≤65 years of age (Treatment B), with Body Mass Index (BMI) >18.5 and <30.0 kg/m2
* Females of childbearing potential must be willing to use a medically acceptable method of birth control throughout the study
* Capable of consent

Exclusion Criteria:

* Any clinically significant abnormality or abnormal laboratory test results found during medical screening
* Positive hepatitis B, hepatitis C, HIV, urine drug screen, urine cotinine test, or alcohol breath test at screening
* History of allergic reactions to cyclobenzaprine, any of the formulation component, or other related drugs
* Use of any drugs known to induce or inhibit hepatic drug metabolism within 30 days prior to the first study drug administration
* Positive pregnancy test at screening
* Clinically significant electrocardiogram (ECG) abnormalities or vital sign abnormalities at screening
* History of significant alcohol or drug abuse within one year prior to screening
* Participation in a clinical trial involving the administration of an investigational or marketed drug within 30 days prior to the first dosing or concomitant participation in an investigational study involving no drug administration
* Use of medication other than topical products without significant systemic absorption and hormonal contraceptives
* Donation of plasma within 7 days prior to dosing, or significant loss of blood within 54 days of dosing.
* Abnormal hemoglobin and hematocrit levels at screening
* Breast-feeding subject
* Presence of dentures, tongue piercings with ongoing use of tongue studs/jewelry, orthodontic braces, or surgical manipulations of the tongue

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2018-04-09 (Actual); Study Completion 2018-04-09 (Actual)

PRIMARY OUTCOMES:
Steady-State Area Under the Plasma Concentration Versus Time Curve (AUC-ss) of TNX-102 SL 5.6 mg versus AMRIX 30 mg | Day 1 to Day 27
  Blood samples are collected from pre-dose on Day 1 up until Day 27 (168 hours post-last dose).
Peak Steady-State Plasma Concentration (Cmax-ss) of TNX-102 SL 5.6 mg versus AMRIX 30 mg | Day 1 to Day 27
  Blood samples are collected from pre-dose on Day 1 up until Day 27 (168 hours post-dose).
Number of Subjects With Treatment-Emergent Adverse Events (TEAEs) of TNX-102 SL 5.6 mg versus AMRIX 30 mg | Day 1 to Day 47
  TEAEs will be collected throughout the study and are summarized descriptively by treatment, relationship, and severity for all subjects dosed.
Peak Steady-State Plasma Concentration (Cmax-ss) of norcyclobenzaprine from TNX-102 SL 5.6 mg versus AMRIX 30 mg | Day 1 to Day 47
  Blood samples are collected from pre-dose on Day 1 up until Day 47 (648 hours post-last dose).

CONTACTS AND LOCATIONS:
Locations (1):
- Quebec City, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided